CLINICAL TRIAL: NCT02064686
Title: EXHALED AIR TEMPERATURE (TAE) AS A MARKER OF AIRWAY INFLAMMATION IN ASTHMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: IIBSP-TAE-2011-145; 09/078/992
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: ASTHMA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAE (No Intervention)
  Interventions: Other: Exhaled breath temperature

INTERVENTIONS:
Other: Exhaled breath temperature

SUMMARY:
The goals : to develop and computerize equipment for measuring ITAE , compare the results with TAEP Itae study the possible relationship between different markers of inflammation: sputum eosinophils , FeNO , the ITAE and TAEP and see the influence spirometry or a bronchodilator in measuring the ITAE .

It has designed a line of work studying the following aspects :

1. Comparison with TAEP ITAE in a group of healthy and stable asthmatics 60 patients , 30 asthma and 30 volunteers .

Two . Study of the relationship between the number of eosinophils in sputum, FeNO , the ITAE and TAEP , 30 patients randomly FeNO , the ITAE and TAEP be measured.

Three . ITAE measurement before and after the spirometry test , 20 patients , in stable phase will be measured before and after the ITAE spirometry .

April . ITAE baseline measurement and after administration of 400 micrograms of salbutamol , 20 patients diagnosed with asthma , phase stable , they measure the ITAE before and fifteen minutes after administration of salbutamol .

May . Measurement in patients Itae a bronchial provocation test with methacholine was performed , 20 patients were measured and baseline Itae after administration of methacholine .

6. Measuring Itae in patients during an asthma exacerbation and stable phase , 20 patients during an exacerbation , the ITAE be measured. Already in clinically stable measurement is repeated.

DETAILED DESCRIPTION:
The goals : to develop and computerize equipment for measuring ITAE , compare the results with TAEP Itae study the possible relationship between different markers of inflammation: sputum eosinophils , FeNO , the ITAE and TAEP and see the influence spirometry or a bronchodilator in measuring the ITAE .

It has designed a line of work studying the following aspects :

1. Comparison with TAEP ITAE in a group of healthy and stable asthmatics 60 patients , 30 asthma and 30 volunteers .

Two . Study of the relationship between the number of eosinophils in sputum, FeNO , the ITAE and TAEP , 30 patients randomly FeNO , the ITAE and TAEP be measured.

Three . ITAE measurement before and after the spirometry test , 20 patients , in stable phase will be measured before and after the ITAE spirometry .

April . ITAE baseline measurement and after administration of 400 micrograms of salbutamol , 20 patients diagnosed with asthma , phase stable , they measure the ITAE before and fifteen minutes after administration of salbutamol .

May . Measurement in patients Itae a bronchial provocation test with methacholine was performed , 20 patients were measured and baseline Itae after administration of methacholine .

6. Measuring Itae in patients during an asthma exacerbation and stable phase , 20 patients during an exacerbation , the ITAE be measured. Already in clinically stable measurement is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with asthma

Exclusion Criteria:

* Patients unable to perform the maneuver the measurement of the TAE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Exhaled Breath Temperature (TAE) As A Marker Of Airway Inflammation In Asthma | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Giner, MSc, Principal Investigator — Hospital de la Sta. Creu i Sant Pau
Locations (1):
- Hospital de la Sta. Creu i Sant Pau, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Paredi P, Kharitonov SA, Barnes PJ. Faster rise of exhaled breath temperature in asthma: a novel marker of airway inflammation? Am J Respir Crit Care Med. 2002 Jan 15;165(2):181-4. doi: 10.1164/ajrccm.165.2.2103053. PMID 11790651
- [Background] Piacentini GL, Bodini A, Zerman L, Costella S, Zanolla L, Peroni DG, Boner AL. Relationship between exhaled air temperature and exhaled nitric oxide in childhood asthma. Eur Respir J. 2002 Jul;20(1):108-11. doi: 10.1183/09031936.02.00237702. PMID 12166556
- [Background] Paredi P, Kharitonov SA, Barnes PJ. Correlation of exhaled breath temperature with bronchial blood flow in asthma. Respir Res. 2005 Feb 10;6(1):15. doi: 10.1186/1465-9921-6-15. PMID 15705206
- [Background] Popov TA, Dunev S, Kralimarkova TZ, Kraeva S, DuBuske LM. Evaluation of a simple, potentially individual device for exhaled breath temperature measurement. Respir Med. 2007 Oct;101(10):2044-50. doi: 10.1016/j.rmed.2007.06.005. Epub 2007 Jul 12. PMID 17624752